CLINICAL TRIAL: NCT05709522
Title: Neurocognitive and Psychosocial Outcomes Among Pediatric Brain Tumor and Blood Cancer Patients Presenting to a Tertiary Care Hospital of Karachi, Pakistan: A Prospective Cohort Study
Brief Title: Neurocognitive and Psychosocial Outcomes Among Pediatric Brain Tumor and Blood Cancer Patients
Acronym: PBT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Nida Zahid, Principal Investigator, Aga Khan University
Other Study IDs: 2021-4859-18168.
Record Dates: First submitted 2021-06-15; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Brain Tumor, Pediatric; Blood Cancer
Keywords: Pediatric Brain tumor; Blood Cancer; Neurocognition; Psychosocial outcomes; Quality of life; depression; socioeconomic burden
MeSH Terms: conditions — Brain Neoplasms; Hematologic Neoplasms; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be stored to assess microRNA and Protein markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric brain tumor patients: The study participants will be 5 to 21 years old children with newly diagnosed brain tumors presenting with any stage, who have not undergone any treatment
  Interventions: Behavioral: Neurocognitive tools
- Blood cancer children: The study participants will be 5 to 21 years old children with newly diagnosed blood cancer presenting with any stage, who have not undergone any treatment
  Interventions: Behavioral: Neurocognitive tools

INTERVENTIONS:
Behavioral: Neurocognitive tools — Neurocognitve and psychological tools
  Other Names: Psychosocial tools

SUMMARY:
This will be the first in-depth study to evaluate pretreatment and 12 months post-treatment, neurocognitive and psychological outcomes of children with brain tumor and blood cancer in Pakistan. The investigators will also determine the socioeconomic burden of pediatric brain tumors in low middle-income region and the association of micro RNA and protein markers with neurocognitive outcomes in PBT and blood cancer children. A prospective cohort study with a follow-up of 12 months at the Aga Khan University Hospital, Karachi, Pakistan and Jinnah postgraduate Medical Centre , Karachi, Pakistan will be conducted. After taking consent/ assent the investigators will recruit 80, 5-21 years old children with newly diagnosed brain tumors presenting with any stage, who have not undergone any treatment. Trained psychologist will assess the neurocognitive outcomes by the Slosson scale, Raven's progressive matrices and Wechsler Intelligence Scale for children (WISC V) and Wechsler Adult Intelligence Scale (WAIS-IV) tools. The Quality of life and depression of the children will be determined by PedQL and Revised Children's Anxiety and Depression Scale (RCADS) and hospital anxiety and depression scale (HADs) respectively . The financial burden of the disease on the family will be measured on a visual analog scale ranging from no burden (0) to very large burden (100) and the parents QoL and disrupted schedule, financial problems, lack of family support, health problems and the impact of caregiving on caregiver's self-esteem will be assessed by Pediatric Quality of Life Inventory PedQl (family module) and Caregiver Reaction Assessment (CRA) tools respectively. The serum micro RNA (mi-21, mi-10b and mi-210) and protein markers (GFAP, NSE and S100β) will be assessed by qRT-PCR and ELISA.

DETAILED DESCRIPTION:
Rationale: The synergy between poverty, socio-cultural, psychosocial and biological risk factors influences neurocognitive outcomes in children. In a LMIC like ours where children are growing up at a disadvantage, it is important the child's future potential and productivity. To the best of the investigators knowledge limited information, there is no data in this area from Pakistan. Data to assess the neurocognitive and psychological outcomes of children during this vulnerable period and to design interventions which may help to improve from this study will be enable the assessment of direction and magnitude of effects, identify high risk children whom would benefit from individual treatment and, with this knowledge, enhance family support Study Design and Site A prospective cohort study with a follow-up of 12 months. The study will be conducted at the Aga Khan University Hospital (AKUH) and Jinnah post graduate Medical Centre (JPMC). The participants will be recruited from the neurosurgery/oncology clinics.

Study Participants The study participants will be 5 to 21 years old children with newly diagnosed brain tumors and blood cancer presenting with any stage, who have not undergone any treatment

Sampling strategy Purposive sampling technique will be used for selecting the participants. The target population, that is, brain tumor and blood cancer children who have not received cancer treatment, will be approached by trained psychologist.

Sample size: With a mean difference of neurocognitive outcome ranging from 15 to 23 and difference of standard deviation ranging from 14 to 27, from pretreatment to 12 months post treatment .And with a mean difference of Quality of life ranging from 9 to 16 and difference of standard deviation ranging from 18 to 19 . With a power of 80% and level of significance of 5%. However, the investigators calculated the sample size using two population mean in order to compare the mean neurocognitive and psychological scores of the two groups. With an anticipated mean difference of 6, a standard deviation of 15 for the two groups, a level of significance of 5%, and power of 80%. Therefore the final sample size will be 80 patients ( 40 pediatric brain tumor patients and 40 blood cancer patients), with a 10% inflation for loss to follow-up

Data collection The children with brain tumor and blood cancer will be recruited from the surgery/ pediatric oncology clinics AKUH. Screening tool will be administered for eligibility of the study participant for the study. The Pediatric Quality of Life Inventory , PedsQL family information form will be completed by the parents that contains demographic information required to calculate Hollingshead socioeconomic status (SES). Information will also be collected on; tumor and treatment related factors, histopathology, family history, nutritional status, consanguinity and perinatal risk factors and molecular expression analysis chart on a structured questionnaire for pediatric brain tumor patients and blood cancer patients

The neurocognitive outcomes of the eligible children will be assessed by a psychologist at baseline i.e., before treatment and 12 months post-treatment. It will be assessed by the Slosson Intelligence tool Revised 3rd edition (SIT-R3) and Raven's Progressive Matrices (RPM).The progressing speed will be assessed by Wechsler Intelligence Scale for children (WISC V) and Wechsler Adult Intelligence Scale (WAIS-IV)

Plan of Analysis Data will be analyzed using STATA version 15. Results will be presented as mean and standard error/ median , interquartile range (IQR) for cognitive outcomes, quality of life (QoL) scores and financial burden scores. Pretreatment and 12 months post treatment scores will be assessed by paired t test/ wilcoxon sign rank test as appropriate. Categorical variables will be reported as frequency and percentages and will be assessed by chi-square/ fisher exact test. Correlation analysis will be preformed to assess relationship of child's neurocognitive outcome scores with QoL scores and child's QoL scores with the parents QoL scores. Unadjusted and adjusted beta coefficient with 95% CI will be reported by using Linear mixed effects models (LMEMs) to determine the association of various independent factors such as child factors (demographic factors), parental factors (educational status, socioeconomic status, prenatal exposure/ infections) , tumor and treatment related factors with the neurocognitive outcomes and QoL. We will adjust for the independent variables and determine the association of factors causing a greater decline in outcomes by multivariable Linear mixed effects models (LMEMs) . Plausible interactions will also be assessed. A p value of < 0.05 will be considered as significant throughout the study

ELIGIBILITY:
Inclusion Criteria:

1. 5-21 years children with brain tumor, presenting with any stage
2. Children residing in Pakistan for at least 3 months.
3. Children accompanied by both or either of the parent
4. Children with basic understanding of English
5. Children and their parents who understand and speak in Urdu
6. Children and their parents who will give assent / consent to participate in the study

Exclusion Criteria:

1. Children who have received any type of treatment for brain tumor and blood cancer
2. Children presenting with recurrence
3. Children with metastatic brain tumor and blood cancer
4. Known cases of any illness leading to psychiatric/neurological illness (e.g. ADHD, autism, schizophrenia) as confirmed by medical records, will be excluded from the study as they may be on medications that might distort the results.
5. Children with physical comorbidities and debilitating disease
6. Children who will loss to follow-up

   -

Ages: 5 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: 5-21 years old pediatric brain tumor and blood cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Neuro-cognitive outcomes | November 2020 to November 2023
  The Verbal component of neurocognition will be assessed by slosson scale.A higher score means a better outcome
Neuro-cognitive outcomes | November 2020 to November 2023
  The non verbal component of neurocognition will be assessed by Raven tool (non verbal) a higher score means good neurocognition
Neuro-cognitive outcomes | November 2020 to November 2023
  The non verbal component i.,e processing speed of neurocognition will be assessed by Wechler scale . A high score means good neurocognition
Quality of life of child | November 2020 to November 2023
  Pediatric Quality of Life Inventory tools ( generic, brain module and cancer module); Score 0-100; higher scores means good Quality of life
Depression and anxiety | November 2020 to November 2023
  Revised Children's Anxiety and Depression Scale and hospital anxiety and depression scale; score 0-141 a higher score mean high depression and anxiety; 0-7 mild depression and anxiety; 8=10 moderate depression and anxiety and 11-21 severe depression and anxiety

SECONDARY OUTCOMES:
Parents health related Quality of life | November 2020 to November 2023
  Pediatric Quality of Life™ Family Impact Module will be used to assess parents quality of life ; a higher score means a good Quality of life
MicroRNA | November 2020 to November 2023
  serum micro RNA (mi-21, mi-10b and mi-210) and will be assessed by qRT-PCR
S100 calcium-binding protein B (S100β) | November 2020 to November 2023
  protein markers S100β will be assessed by ELISA
Neurons and peripheral neuroendocrine cells (NSE) | November 2020 to November 2023
  protein markers NSE will be assessed by ELISA
Glial fibrillary acidic protein (GFAP) | November 2020 to November 2023
  protein markers GFAP will be assessed by ELISA
financial burden of the disease on the family; | November 2020 to November 2023
  visual analog scale ranging from no burden (0) to very large burden (100). high score and means higher burden of the disease
Care giver Reaction scale Caregiver Reaction Assessment (CRA) tool ) | November 2020 to November 2023
  The questionnaire consists of 24 items measuring five subscales: impact on disrupted schedule, financial problems, lack of family support, health problems and impact on self-esteem. Caregivers have to indicate their level of agreement using a 5-point Likert-type Scale ranging from 1 (strongly disagree) to 5 (strongly agree). For each subscale, a score is calculated by taking the average of the items. Higher scores indicate a greater impact (either beneficial or detrimental).

CONTACTS AND LOCATIONS:
Locations (1):
- Nida Zahid, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zahid N, Enam SA, Martensson T, Azam I, Mushtaq N, Moochhala M, Javed F, Kausar F, Hasan A, Rehman L, Mughal MN, Altaf S, Kirmani S, Brown N. Predictors of neurocognition outcomes in children and young people with primary brain tumor presenting to tertiary care hospitals of Karachi, Pakistan: a prospective cohort study. Childs Nerv Syst. 2024 Jun;40(6):1707-1719. doi: 10.1007/s00381-024-06306-x. Epub 2024 Feb 16. PMID 38363314